CLINICAL TRIAL: NCT06773416
Title: Treating Sleep Apnea to Improve Cognitive Function, Alzheimer's Disease Pathology, and Astrocyte Activation in Older Adults With Cognitive Impairment: A Multi-Centre Randomized Controlled Trial
Brief Title: CPAP Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Baycrest (Other); University Health Network, Toronto (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTO 5040; BH-10967 (Other Grant/Funding Number: Weston Family Foundation)
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Obstructive Sleep Apnea (OSA); Mild Cognitive Impairment (MCI); Cognitive Decline Prevention in Pre-frail Older Adults
Keywords: Obstructive Sleep Apnea; Cognitive Decline; CPAP Therapy; Mild Cognitive Impairment; Dementia Prevention; Sleep Education; Brain Health; Cognitive Function; Randomized Controlled Trial; CPAP Adherence; Older Adults; Alzheimer's Disease
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two groups: Group 1 is an Early CPAP group and Group 2 is a Later CPAP group. Group 1 begins CPAP therapy alongside web-based sleep education from baseline whereas Group 2 starts CPAP therapy after 4 months of web-based sleep education, similar to current clinical practices.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (Early CPAP group) (Experimental): Participant will receive a study-provided CPAP device at their baseline visit, with settings set by one of the study sleep medicine physicians according to current clinical practice parameters. Participant will undergo an in-person mask fitting and then will be supported by a study sleep technologist with extensive clinical experience with CPAP who will contact the participant by telephone or video call at set intervals. Masks, tubing, chin straps, and other equipment necessary to optimize CPAP adherence will be provided by the study. Adherence will be monitored through downloads from the CPAP device. Participant will be asked to use CPAP nightly during their participation in this study. Participant will simultaneously participate in web-based sleep education through the Brain Health Pro (BHP) platform; a formal educational program designed to increase dementia literacy, foster engagement, and convey best available evidence for lifestyle changes that can mitigate dementia risk.
  Interventions: Combination Product: CPAP Therapy Combined with Web-Based Sleep Education for Cognitive and Sleep Health
- Group 2 (Later CPAP group) (Active Comparator): Participant will receive the web-based sleep educational intervention first for 4 months. Participant will then receive a study-supplied CPAP device with settings set by one of the study sleep medicine physicians according to current clinical practice parameters. Participant will undergo an in-person mask fitting and will be supported by a study sleep technologist with extensive clinical experience with CPAP who will contact the participant by telephone or video call at set intervals. Equipment necessary to optimize CPAP adherence will be provided. Adherence will be monitored through downloads from the CPAP device. Participant will be asked to use CPAP nightly throughout their participation. Participant will simultaneously participate in web-based sleep education through the Brain Health Pro platform; a formal educational program designed to increase dementia literacy, foster engagement and convey best available evidence for lifestyle changes that can mitigate dementia risk.
  Interventions: Combination Product: Delayed CPAP Therapy Combined with Web-Based Sleep Education for Cognitive and Sleep Health

INTERVENTIONS:
Combination Product: CPAP Therapy Combined with Web-Based Sleep Education for Cognitive and Sleep Health — Participants in Group 1 will receive CPAP therapy immediately upon enrollment alongside web-based sleep education through the Brain Health Pro (BHP) platform. The CPAP intervention includes a study-provided auto-titrating device, in-person mask fitting, and ongoing support from a study sleep technologist. Adherence will be monitored via remote data uploads. The BHP platform is a 45-week web-based formal educational program program designed to increase dementia literacy, foster engagement, and convey best available evidence for lifestyle changes that can mitigate dementia risk. This combined approach ensures simultaneous initiation of CPAP and educational reinforcement to optimize adherence and cognitive outcomes.
  Arms: Group 1 (Early CPAP group)
Combination Product: Delayed CPAP Therapy Combined with Web-Based Sleep Education for Cognitive and Sleep Health — Participants in Group 2 will begin with 4 months of BHP web-based sleep education before adding CPAP therapy for the remaining 4 months. CPAP setup and support are identical to the Early CPAP group. Participants in Group 2 will experience procedure similar to current clinical practices.
  Arms: Group 2 (Later CPAP group)

SUMMARY:
The overall goal of this randomized controlled trial is to test the hypothesis that in older adults with mild cognitive impairment (MCI) and previously untreated obstructive sleep apnea (OSA), 4 months of web-based sleep education and continuous positive airway pressure (CPAP) will improve cognitive function more than web-based sleep education alone. Secondarily, this trial will test the hypothesis that 8 months of CPAP will improve cognitive function more than 4 months of CPAP. Moreover, treating OSA with CPAP can improve cognitive function and reduce Alzheimer's disease-related brain changes in older adults with MCI.

This study will compare an Early CPAP Group who will receive CPAP and sleep education simultaneously for 8 months upon enrollment to a Later CPAP Group who will first receive sleep education for 4 months followed by CPAP and sleep education for the next 4 months to test if early treatment is more beneficial.

Participants will:

1. Complete web-based sleep education modules through the Brain Health Pro (BHP) platform
2. Undergo CPAP therapy, including in-person mask fitting and regular monitoring alongside a study sleep technologist

At 0 months, 4 months, and 8 months, participants will participate in cognitive assessments, provide blood samples, use wearable devices to measure sleep patterns and physiology, and complete a 1-hr MRI (0 months and 4 months only).

DETAILED DESCRIPTION:
This clinical study is a single-blinded, randomized controlled trial of 206 adults designed to evaluate the impact of CPAP therapy on cognitive function and Alzheimer's disease-related pathology in older adults with MCI and untreated OSA. Participants will be randomized into two groups: the first group receiving CPAP treatment alongside sleep education upon enrollment for 8 months (Early CPAP group) and the other beginning CPAP treatment after 4 months of sleep education (Later CPAP group).

1. Early CPAP Group: Participants randomized to this group will start BHP-sleep and CPAP simultaneously and continue both for 8 months. BHP-sleep consists of the sleep modules of the Canadian Consortium on Neurodegeneration in Aging's (CCNA) online Brain Health PRO platform covering sleep physiology, healthy sleep habits, and information about sleep disorders like sleep apnea. Participants will receive a study-provided auto-titrating CPAP device, with settings set by one of the study sleep medicine physicians according to current clinical practice parameters. Participants will undergo an in-person mask fitting, and then will be supported by a sleep technologist with extensive clinical experience with CPAP.
2. Later CPAP Group: Participants randomized to this group will start BHP-sleep without CPAP for first 4 months, followed by BHP-sleep and CPAP simultaneously for remaining 4 months of participation.

Participants in both groups will register at baseline for the web-based sleep education through the Brain Health Pro (BHP) platform; a 45-week, multidomain, web-based formal educational program designed to increase dementia literacy, foster engagement, and convey best available evidence for lifestyle changes that can mitigate dementia risk. This protocol will utilize the sleep modules of the BHP platform covering sleep physiology, healthy sleep habits, and information about sleep disorders like sleep apnea.

This trial will assess cognitive function primarily using the Symbol Digit Modalities Test (SDMT); a test of speeded executive function that is predictive of clinically significant improvement in patients with MCI, alongside additional cognitive measures that supplement the primary outcome of this study will be: attention and executive function (Trail Making Test A & B), working memory (Digit Span and Letter-Number Sequencing), verbal learning and memory (Hopkins Verbal Learning Test), and severity of cognitive impairment (Alzheimer's Disease Assessment Scale - Cognitive Subscale; ADAS-Cog-13).

This trial will also quantify brain perivascular spaces (PVS) volume and structural changes, plasma glial fibrillary acidic protein (GFAP) and plasma pTau-181.

This trial will also aim to identify features of sleep physiology that mediate the impact of CPAP on cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained and signed
* Age >55
* MCI: Participants will undergo a video-based screening, including a clinical interview, Logical Memory II, MoCA, and Lawton-Brody Instrumental Activities of Daily Living Scale Score. A participant will be considered to have MCI if they have: 1) MoCA score of 13-24 and Logical Memory II Score ≤ 8 (&=16 years of education), ≤ 4 (8-15 years of education) or ≤ 2 (0-7 years of education) and Lawton-Brody IADL Score >14/23 and do not meet DSM IV criteria for dementia and have a change in self-perceived cognition from previous
* Moderate-severe OSA: Participants who screen positive for MCI will be mailed an at-home sleep apnea testing device. Participants with ODI≥5 will undergo in-lab polysomnography (PSG) for confirmation and characterization of sleep apnea. A participant will be considered to have moderate-severe OSA if they have on PSG: AHI>15, and ODI>10, and central apneas<10% of all apneas, and periodic limb movement index <15.

Exclusion Criteria:

* drowsiness-related driving accidents or near misses in the past 12 months
* drives as their primary occupation
* unable to complete cognitive evaluation in English
* unable to participate in video-based cognitive assessment
* not a resident of Ontario
* contraindications to MRI
* contraindications to CPAP or unwilling to start CPAP
* no available study partner to support CPAP
* previously treated for sleep apnea
* clinically significant insomnia (ISI > 15), restless legs syndrome, or shift work
* taking disease modifying agents for MCI

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in Symbol Digit Modalities Test (SDMT) | From Week 0 to Week 32
  The SDMT is a test of speeded executive function that is predictive of clinically significant improvement in patients with MCI with a well-defined minimal clinically significant change and that is responsive to CPAP in observational studies. Additional cognitive measures that supplement the primary outcome of this study will be: attention and executive function (Trail Making Test A & B), working memory (Digit Span and Letter-Number Sequencing), verbal learning and memory (Hopkins Verbal Learning Test), and severity of cognitive impairment (Alzheimer's Disease Assessment Scale - Cognitive Subscale; ADAS-Cog-13).

SECONDARY OUTCOMES:
Vascular Risk Factors and AD-biomarkers | From Week 0 to Week 32
  Quantification of plasma pTau181 (AD pathology) using ptau-181 V2.1 Advantage Assay and GFAP (astrocyte activation) using the GFAP discovery assay.
  Blood levels of various fats, sugars and proteins (such as cholesterol or glucose) will be assessed.
  Sleep physiology will be assessed using wearable sensors: at-home sleep apnea testing apparatus (for oximetry metrics including AHI, ODI, mean SpO2, hypoxia burden, and time with O2<92%), EEG headband (sleep staging, including % slow wave sleep, % REM sleep, total EEG sleep time, and NREM slow wave power), and wrist-worn accelerometry (for total sleep time and sleep fragmentation).
MRI | From Week 0 to Week 16
  Participants will undergo MRI using the Canadian Dementia Imaging protocol consisting of a 3D T1, interleaved 3mm PD/T2, 3D FLAIR, T2*, DTI, and resting state BOLD. Perivascular spaces and white matter hyperintensities will be quantified with the SynthSegCSVD algorithm developed and validated in our laboratory, a robust neural network based tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hedner J, White DP, Malhotra A, Herscovici S, Pittman SD, Zou D, Grote L, Pillar G. Sleep staging based on autonomic signals: a multi-center validation study. J Clin Sleep Med. 2011 Jun 15;7(3):301-6. doi: 10.5664/JCSM.1078. PMID 21677901
- [Background] Onder NS, Akpinar ME, Yigit O, Gor AP. Watch peripheral arterial tonometry in the diagnosis of obstructive sleep apnea: influence of aging. Laryngoscope. 2012 Jun;122(6):1409-14. doi: 10.1002/lary.23233. Epub 2012 Apr 20. PMID 22522750
- [Background] Crowley KE, Rajaratnam SM, Shea SA, Epstein LJ, Czeisler CA, Lockley SW; Harvard Work Hours, Health and Safety Group. Evaluation of a single-channel nasal pressure device to assess obstructive sleep apnea risk in laboratory and home environments. J Clin Sleep Med. 2013 Feb 1;9(2):109-16. doi: 10.5664/jcsm.2400. PMID 23372462
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Benedict RHB, Schretlen D, Groninger L, & Brandt J (1998). Hopkins Verbal Learning Test - Revised: Normative Data and Analysis of Inter-Form and Test-Retest Reliability. The Clincal Neuropsychologist, 12(1), 43-55.
- [Background] Wechsler D. The Psychological Corporation; 1997. WMS-III Administration and Scoring Manual.
- [Background] Esther Strauss, O. S. (1998). Trail Making Tests. New York, Oxford University Press.
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] DOPPELT JE, WALLACE WL. Standardization of the Wechsler adult intelligence scale for older persons. J Abnorm Psychol. 1955 Sep;51(2):312-30. doi: 10.1037/h0044391. No abstract available. PMID 13263050
- [Background] Chapman JE, Cadilhac DA, Gardner B, Ponsford J, Bhalla R, Stolwyk RJ. Comparing face-to-face and videoconference completion of the Montreal Cognitive Assessment (MoCA) in community-based survivors of stroke. J Telemed Telecare. 2021 Sep;27(8):484-492. doi: 10.1177/1357633X19890788. Epub 2019 Dec 9. PMID 31813317
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Boeve BF, Molano JR, Ferman TJ, Smith GE, Lin SC, Bieniek K, Haidar W, Tippmann-Peikert M, Knopman DS, Graff-Radford NR, Lucas JA, Petersen RC, Silber MH. Validation of the Mayo Sleep Questionnaire to screen for REM sleep behavior disorder in an aging and dementia cohort. Sleep Med. 2011 May;12(5):445-53. doi: 10.1016/j.sleep.2010.12.009. Epub 2011 Feb 23. PMID 21349763
- [Background] Allen RP, Burchell BJ, MacDonald B, Hening WA, Earley CJ. Validation of the self-completed Cambridge-Hopkins questionnaire (CH-RLSq) for ascertainment of restless legs syndrome (RLS) in a population survey. Sleep Med. 2009 Dec;10(10):1097-100. doi: 10.1016/j.sleep.2008.10.007. Epub 2009 Feb 4. PMID 19195928
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Chung F, Abdullah HR, Liao P. STOP-Bang Questionnaire: A Practical Approach to Screen for Obstructive Sleep Apnea. Chest. 2016 Mar;149(3):631-8. doi: 10.1378/chest.15-0903. Epub 2016 Jan 12. PMID 26378880
- [Background] Lim AS, Yu L, Kowgier M, Schneider JA, Buchman AS, Bennett DA. Modification of the relationship of the apolipoprotein E epsilon4 allele to the risk of Alzheimer disease and neurofibrillary tangle density by sleep. JAMA Neurol. 2013 Dec;70(12):1544-51. doi: 10.1001/jamaneurol.2013.4215. PMID 24145819
- [Background] Feldman HH, Belleville S, Nygaard HB, Montero-Odasso M, Durant J, Lupo JL, Revta C, Chan S, Cuesta M, Slack PJ, Winer S, Brewster PWH, Hofer SM, Lim A, Centen A, Jacobs DM, Anderson ND, Walker JD, Speechley MR, Zou GY, Chertkow H. Protocol for the Brain Health Support Program Study of the Canadian Therapeutic Platform Trial for Multidomain Interventions to Prevent Dementia (CAN-THUMBS UP): A Prospective 12-Month Intervention Study. J Prev Alzheimers Dis. 2023;10(4):875-885. doi: 10.14283/jpad.2023.65. PMID 37874110
- [Background] Richards KC, Lozano AJ, Morris J, Moelter ST, Ji W, Vallabhaneni V, Wang Y, Chi L, Davis EM, Cheng C, Aguilar V, Khan S, Sankhavaram M, Hanlon AL, Wolk DA, Gooneratne N. Predictors of Adherence to Continuous Positive Airway Pressure in Older Adults With Apnea and Amnestic Mild Cognitive Impairment. J Gerontol A Biol Sci Med Sci. 2023 Oct 9;78(10):1861-1870. doi: 10.1093/gerona/glad099. PMID 37021413
- [Background] Morgenthaler TI, Aurora RN, Brown T, Zak R, Alessi C, Boehlecke B, Chesson AL Jr, Friedman L, Kapur V, Maganti R, Owens J, Pancer J, Swick TJ; Standards of Practice Committee of the AASM; American Academy of Sleep Medicine. Practice parameters for the use of autotitrating continuous positive airway pressure devices for titrating pressures and treating adult patients with obstructive sleep apnea syndrome: an update for 2007. An American Academy of Sleep Medicine report. Sleep. 2008 Jan;31(1):141-7. doi: 10.1093/sleep/31.1.141. PMID 18220088
- [Background] Yalamanchali S, Farajian V, Hamilton C, Pott TR, Samuelson CG, Friedman M. Diagnosis of obstructive sleep apnea by peripheral arterial tonometry: meta-analysis. JAMA Otolaryngol Head Neck Surg. 2013 Dec;139(12):1343-50. doi: 10.1001/jamaoto.2013.5338. PMID 24158564
- [Background] Chatterjee P, Dore V, Pedrini S, Krishnadas N, Thota R, Bourgeat P, Ikonomovic MD, Rainey-Smith SR, Burnham SC, Fowler C, Taddei K, Mulligan R, Ames D, Masters CL, Fripp J, Rowe CC, Martins RN, Villemagne VL; The AIBL Research Group. Plasma Glial Fibrillary Acidic Protein Is Associated with 18F-SMBT-1 PET: Two Putative Astrocyte Reactivity Biomarkers for Alzheimer's Disease. J Alzheimers Dis. 2023;92(2):615-628. doi: 10.3233/JAD-220908. PMID 36776057
- [Background] Mielke MM, Hagen CE, Xu J, Chai X, Vemuri P, Lowe VJ, Airey DC, Knopman DS, Roberts RO, Machulda MM, Jack CR Jr, Petersen RC, Dage JL. Plasma phospho-tau181 increases with Alzheimer's disease clinical severity and is associated with tau- and amyloid-positron emission tomography. Alzheimers Dement. 2018 Aug;14(8):989-997. doi: 10.1016/j.jalz.2018.02.013. Epub 2018 Apr 5. PMID 29626426
- [Background] Jack CR, Wiste HJ, Algeciras-Schimnich A, Figdore DJ, Schwarz CG, Lowe VJ, Ramanan VK, Vemuri P, Mielke MM, Knopman DS, Graff-Radford J, Boeve BF, Kantarci K, Cogswell PM, Senjem ML, Gunter JL, Therneau TM, Petersen RC. Predicting amyloid PET and tau PET stages with plasma biomarkers. Brain. 2023 May 2;146(5):2029-2044. doi: 10.1093/brain/awad042. PMID 36789483
- [Background] Richards KC, Gooneratne N, Dicicco B, Hanlon A, Moelter S, Onen F, Wang Y, Sawyer A, Weaver T, Lozano A, Carter P, Johnson J. CPAP Adherence May Slow 1-Year Cognitive Decline in Older Adults with Mild Cognitive Impairment and Apnea. J Am Geriatr Soc. 2019 Mar;67(3):558-564. doi: 10.1111/jgs.15758. Epub 2019 Feb 6. PMID 30724333
- [Background] Borland E, Edgar C, Stomrud E, Cullen N, Hansson O, Palmqvist S. Clinically Relevant Changes for Cognitive Outcomes in Preclinical and Prodromal Cognitive Stages: Implications for Clinical Alzheimer Trials. Neurology. 2022 Sep 13;99(11):e1142-e1153. doi: 10.1212/WNL.0000000000200817. Epub 2022 Jul 14. PMID 35835560
- [Background] Yaffe K, Laffan AM, Harrison SL, Redline S, Spira AP, Ensrud KE, Ancoli-Israel S, Stone KL. Sleep-disordered breathing, hypoxia, and risk of mild cognitive impairment and dementia in older women. JAMA. 2011 Aug 10;306(6):613-9. doi: 10.1001/jama.2011.1115. PMID 21828324

DOCUMENTS (2):
  • Study Protocol (2024-11-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT06773416/Prot_000.pdf
  • Informed Consent Form (2024-11-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT06773416/ICF_001.pdf